CLINICAL TRIAL: NCT04475068
Title: Feasibility and Physiological Effects of a Postural Recruitment Maneuver in Patients With Acute Respiratory Distress Syndrome Due to COVID-19 Infection
Brief Title: Postural Recruitment Maneuver in Patients With Acute Respiratory Distress Syndrome Due to COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Hospital Nacional Edgardo Rebagliati Martins (Other)
Collaborators: Universidad de Piura (Unknown)
Responsible Party: Principal Investigator, Rollin Roldán, Principal investigator, Hospital Nacional Edgardo Rebagliati Martins
Other Study IDs: HNEdgardoRebagliatiMartins
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Sars-CoV2; ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate to severe ARDS patients due to COVID-19 infection: Mechanically ventilated patients with moderate to severe ARDS due to COVID-19 infection admitted to the COVID Intensive Care Unit of Rebagliati Hospital.
  Interventions: Procedure: Lateral Position (left and right lateral decubitus)

INTERVENTIONS:
Procedure: Lateral Position (left and right lateral decubitus) — Prior to initiating the protocol, patients will be sedated deeply with sedatives and opioids and paralyzed. Patients will be evaluated in 5 positions sequentially: 1) Supine 2) Left lateral 3) Supine 4) Right lateral 5) Supine. The side with the least ventilation evaluated by EIT will define which side will start the sequence. Each step will last 30 minutes. Aeration measured by Electric Impedance Tomography (EIT) and lung ultrasound, distribution of the lung ventilation and perfusion measured by EIT, ventilator and hemodynamic parameters, esophageal pressure, and blood gas analysis will be recorded at the end of each step. Continuous monitoring of blood pressure, heart rate and saturation of arterial blood (SpO2) will be carried out during all steps of the protocol to assess the tolerance to the procedure.

SUMMARY:
The purpose of this study is to evaluate if a postural recruitment maneuver (PRM) improves the aeration and distribution of lung ventilation in patients with Acute Respiratory Distress Syndrome (ARDS) caused by COVID-19 infection; without the need to reach high airway pressures as in the standard lung recruitment maneuver and / or place the patient in prone position. This strategy could be particularly useful in the context of a major health emergency in centers with limited resources.

DETAILED DESCRIPTION:
The PRM is based on the known effect of gravity on transpulmonary pressure (PL). Two principles explain its mechanism of action: 1) the first indicates that atelectasis and poorly ventilated areas of the lung can improve their aeration by putting the lung in the highest position. Opposite lateral decubitus causes that upper lung to have a higher PL and allow a recruiting effect at moderate airway pressures. 2) The second principle is based on Laplace's Law and postulates that once the upper lung is recruited, it remains without lung collapse if a sufficient level of positive end-expiratory pressure (PEEP) is applied. Based on these two precepts, PRM consists of sequentially moving the patient from the supine to the left lateral decubitus to recover the aeration of the right lung. After that, the patient is placed in the right lateral position to recruit the left lung; keeping the right lung without collapse by continuous use of PEEP. Finally, the patient returns to the supine position looking for an improvement in the distribution of ventilation and global pulmonary aeration, with a subsequent improvement in gas exchange and pulmonary mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients with moderate-to-severe ARDS as per the Berlin definition
* Infection due to COVID-19
* Body mass index (BMI) ≤ 35 kg /m^2.

Exclusion Criteria:

* Contraindication for EIT monitoring

  1. Unstable spine or pelvic fractures
  2. Pacemaker, automatic implantable cardioverter defibrillator
  3. Skin lesions between the 4th and 5th ribs where the EIT belt is worn
* Pregnancy
* Major hemodynamic instability::

  1. Mean arterial pressure lower than 60 mm Hg despite adequate fluid resuscitation and use of vasopressors.
  2. FC> 120 or <60 per minute
  3. Presence of uncontrolled arrhythmias.
* More than 1 week of mechanical ventilation
* Failure of more than 2 extrapulmonary organs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This physiological study will enroll 12 adult ARDS patients admitted to the COVID Intensive Care Unit of Rebagliati Hospital. Informed consent will be obtained from the patient or legally authorized substitute decision maker.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Effects of a postural recruitment maneuver in lung aeration | Through study completion (up to 24 hours)
  Lung aeration measured by ultrasound reaeration score, ranges from 0 (all regions are well aerated) to 36 (all regions are consolidated).
Effects of a postural recruitment maneuver in distribution of ventilation | Through study completion (up to 24 hours)
  Distribution of ventilation measured by EIT (distribution and changes in the impedance in AU, arbitray units)
Effects of a postural recruitment maneuver in gas exchange | Through study completion (up to 24 hours)
  Gas exchange measured by blood gas analysis (PaO2, PaCO2, in mmHg) and capnography (end-tidal CO2, in mmHg)
Effects of a postural recruitment maneuver in respiratory mechanics | Through study completion (up to 24 hours)
  Respiratory mechanics measured by esophageal balloon (esophageal pressure, transpulmonary pressure, in cmH2O)
Effects of a postural recruitment maneuver in hemodynamic | Through study completion (up to 24 hours)
  Hemodynamic data measured by invasive arterial monitoring (mean arterial pressure, in mmHg)

SECONDARY OUTCOMES:
Feasibility of a postural recruitment maneuver | Through study completion (up to 24 hours)
  Oxigenatory tolerance evaluated with pulse oximeter (arterial oxygen saturation, in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Rollin Roldán, MD, Principal Investigator — Hospital Nacional Edgardo Rebagliati Martins
Locations (1):
- Hospital Rebagliati, Jesús María, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roldan R, Rodriguez S, Barriga F, Tucci M, Victor M, Alcala G, Villamonte R, Suarez-Sipmann F, Amato M, Brochard L, Tusman G. Sequential lateral positioning as a new lung recruitment maneuver: an exploratory study in early mechanically ventilated Covid-19 ARDS patients. Ann Intensive Care. 2022 Feb 12;12(1):13. doi: 10.1186/s13613-022-00988-9. PMID 35150355